CLINICAL TRIAL: NCT03339466
Title: A Pilot Study of Inspiratory Muscle Function and the Effects of Inspiratory Muscle Training in Subjects With Fontan Physiology
Brief Title: Inspiratory Muscle Therapy in Subjects With Fontan Circulations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Priya Pillutla, Physician Specialist, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30799-01
Record Dates: First submitted 2017-10-18; First posted 2017-11-13 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Single-ventricle
MeSH Terms: conditions — Univentricular Heart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm - Inspiratory Muscle Training (Experimental): Single arm study. All subjects will perform 6-8 weeks of inspiratory muscle therapy with cardiopulmonary stress test (both standard and constant work rate) before and after intervention.
  Interventions: Device: Inspiratory muscle therapy

INTERVENTIONS:
Device: Inspiratory muscle therapy — 6 weeks of inspiratory muscle therapy
  Other Names: No other interventions. Subjects will serve as their own control; single arm study.

SUMMARY:
Individuals who have undergone the Fontan procedure are uniquely dependent upon respiratory mechanics to support pulmonary blood flow (PBF). The investigators hypothesized that enhanced respiratory muscle function via inspiratory muscle training (IMT) would improve performance on cardiopulmonary exercise stress testing (CPET).

DETAILED DESCRIPTION:
Adult Fontan subjects were recruited from 2 academic medical centers. Following characterization of pulmonary function and functional class, CPET was performed using incremental and constant work rate protocols. Subjects performed 6-8 weeks of IMT using a handheld inspiratory loading device (Threshold®, Philips); both exercise tests were then repeated. Patient-centered outcome data were collected before and after IMT (RAND-36 assessment and New York Heart Association (NYHA) functional class).

ELIGIBILITY:
Inclusion Criteria:

Single ventricle physiology status post Fontan palliation

Exclusion Criteria:

* The presence of a sub-pulmonary ventricle
* Pregnancy or any contraindication to stress testing (e.g., uncontrolled symptomatic arrhythmia, severe systemic ventricular outflow tract obstruction or uncontrolled symptomatic heart failure).
* Height less than 4'11" due to limitations of the cycle ergometer.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-01-29 (Actual); Primary Completion 2016-08-24 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Exercise parameters | 6-8 weeks
  Peak VO2 and endurance time are the primary outcome measures

IPD SHARING:
Plan to Share IPD: Undecided